CLINICAL TRIAL: NCT00500812
Title: A Phase I/IIa Dose-Ranging Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BA-210 and the Neurological Status of Patients Following Administration of a Single Extradural Application of Cethrin During Surgery for Acute Thoracic and Cervical Spinal Cord Injury
Brief Title: A Safety Study for Cethrin (BA-210) in the Treatment of Acute Thoracic and Cervical Spinal Cord Injuries
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA-210-101; NCT00104221 (obsolete NCT alias)
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2012-05

CONDITIONS: Spinal Cord Injury
Keywords: biologic drug; transport sequence; rho; spinal cord injury; paralysis; paraplegia; tetraplegia; quadraplegia; trauma; nervous system; fibrin sealant; neurosurgery
MeSH Terms: conditions — Spinal Cord Injuries; Night Blindness, Congenital Stationary, Autosomal Dominant 1; Paralysis; Paraplegia; Quadriplegia; Wounds and Injuries; Neurologic Manifestations | interventions — exoenzyme C3, Clostridium botulinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 0.3 mg (Experimental): Subjects Receiving 0.3 mg Cethrin
  Interventions: Drug: Cethrin
- 1 mg (Experimental): Subjects receiving 1 mg Cethrin
  Interventions: Drug: Cethrin
- 3 mg (Experimental): Subjects receiving 3 mg Cethrin
  Interventions: Drug: Cethrin
- 6 mg (Experimental): Subjects receiving 6 mg Cethrin
  Interventions: Drug: Cethrin
- 9 mg (Experimental): Subjects receiving 9 mg Cethrin
  Interventions: Drug: Cethrin

INTERVENTIONS:
Drug: Cethrin
  Other Names: (BA-210)

SUMMARY:
This trial is a multi-center, open-label, dose-escalation study designed to evaluate the safety, tolerability and pharmacokinetics of Cethrin in two types of spinal cord injury patients: those with a complete cervical injury or a complete thoracic injury. Dose levels from 0.3 mg - 9 mg of Cethrin will be administered.

ELIGIBILITY:
Inclusion Criteria:

Patients will be enrolled in this study only if they meet all of the following criteria:

* Informed Consent Form signed by the patient or patient's legal representative.
* Male or female, aged 16-70 years, inclusive.
* For Group 1, patients with acute thoracic (T2-T12) spinal cord injury; for Group 2, patients with acute cervical (C4-T1) spinal cord injury. The site of surgery should be able to accommodate a minimum volume of 2 mL of fibrin sealant.
* Scheduled to undergo spinal decompression surgery or other interventional spinal surgery (e.g., fixation) within 7 days of injury.
* ASIA Impairment Scale grade of A (complete, no motor or sensory function present in the sacral segment) as assessed within 12 hours before surgery.
* Able to communicate effectively to obtain informed consent and to ensure neurological examination.

Exclusion Criteria:

Patients will not be enrolled in this study if they meet one of the following criteria:

* Use of any experimental drug, or participation in any clinical trial, within 30 days prior to surgery.
* History of adverse reaction to fibrin sealant.
* History of hypersensitivity to bovine products.
* Any medical condition that may interfere with the ASIA assessments.
* Clinically significant neurological, cardiac, respiratory, hepatic, or renal disease or malignancy.
* Hemophilia or other bleeding abnormality as defined by:

  * Platelet level lower than 100 X 109/L
  * Activated partial thromboplastin time or international normalized ratio higher than the upper limit of normal
  * Baseline hematocrit lower than 0.25
* Gunshot wound as the presenting injury, or any evidence of transecting injury to the spinal cord (e.g., by stab wound).
* Cognitive impairment which may preclude accurate neurological assessments (e.g. traumatic head injury with GCS of less than or equal to 14).
* Ankylosing Spondylitis.
* Diabetes mellitus requiring insulin therapy.
* Known immunodeficiency, including Acquired Immune Deficiency Syndrome or use of immunosuppressive or cancer chemotherapeutic drugs.
* Pregnancy or breastfeeding during the study. A serum pregnancy test will be performed at Screening for female patients of childbearing potential. In addition, patients who are considered likely to be pregnant may be excluded at th Investigator's discretion.
* Any condition or situation likely to cause the patient to be unable or unwilling to participate in study procedures or participate in all scheduled study assessments, including follow up through Month 6.
* Any condition likely to result in the patient's death within the next 6 Months.
* Any other condition that, in the opinion of the Investigator, would preclude the patient's participation in the study.
* Previous participation in this study.
* Use of intravenous heparin in previous 48 hours, thrombolytics and/or aspirin containing products in the previous 10 days.
* Non-traumatic causes of spinal cord injury (e.g. transverse myelitis, acute disc herniation, etc…).

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-02; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary goal of this study is to determine the safety and tolerability of Cethrin when administered in conjunction with fibrin sealant to the dura mater of the spinal cord. | Prestudy, 24-72 hrs, 6 weeks, 3, 6 & 12 months

SECONDARY OUTCOMES:
Efficacy by AIS | Pre-study, 24-72 hrs, 6 weeks, 3, 6 & 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Fehlings, MD, PhD, FRCSC, FACS, Principal Investigator — Univestity Health Network, Toronto Western
Locations (8):
- United States (5):
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - University of Cincinnati Mayfield Clinic and Spine Institute, Cincinnati, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Univ.of Virginia Health System, Charlottesville, Virginia
  - University of Washington Harborview Medical Center, Seattle, Washington
- Canada (3):
  - Sunnybrooke Health Sciences Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec

REFERENCES:
- [Result] McKerracher L, Anderson KD. Analysis of recruitment and outcomes in the phase I/IIa Cethrin clinical trial for acute spinal cord injury. J Neurotrauma. 2013 Nov 1;30(21):1795-804. doi: 10.1089/neu.2013.2909. Epub 2013 Oct 1. PMID 23844986
- [Result] Fehlings MG, Theodore N, Harrop J, Maurais G, Kuntz C, Shaffrey CI, Kwon BK, Chapman J, Yee A, Tighe A, McKerracher L. A phase I/IIa clinical trial of a recombinant Rho protein antagonist in acute spinal cord injury. J Neurotrauma. 2011 May;28(5):787-96. doi: 10.1089/neu.2011.1765. PMID 21381984
- See also: Sponsor — http://www.bioaxonebio.com
- See also: Publication — http://www.ncbi.nlm.nih.gov/pubmed?term=mckerracher%20Fehlings